CLINICAL TRIAL: NCT04108611
Title: Role of Online Hemodiafiltration With Endogenous Reinfusion in Treatment of Systemic Lupus Erythematosus Activity Resistant to Conventional Therapy
Brief Title: Immune Adsorption Role in Treatment of Resistant Lupus
Acronym: HFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Mohamed Ahmed El ghiriani (Other)
Responsible Party: Sponsor-Investigator, Dr. Mohamed Ahmed El ghiriani, PhD student, Faculty of medicine, Alexandria university, Egypt, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PhD MElghiriani
Record Dates: First submitted 2019-09-24; First posted 2019-09-30 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Systemic Lupus
Keywords: hemodiafiltration with endogenous re infusion; immune adsorption In Lupus nephritis
MeSH Terms: interventions — Hemodiafiltration

STUDY DESIGN:
Intervention Model Description: Role of online hemodiafiltration with endogenous re infusion in treatment of systemic lupus erythematosus activity resistant to conventional therapy
Masking Description: Patients will not be masked as hemodiafiltration with endogenous re infusion must be observed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- systemic lupus in activity (Experimental): Sixty systemic lupus patients in activity will receive conventional therapy (47 patient as cases 1) and immunadsortion (13 patients as cases 2) will be provided to the non responders
  Interventions: Procedure: hemodiafiltration with endogenous re infusion (HFR)
- Control group 30 subjects (Other): controls 1 (20 healthy volunteers, controls 2 (10 patients with glomerular diseases other than lupus) will do routine laboratory investigations
  Interventions: Procedure: hemodiafiltration with endogenous re infusion (HFR)

INTERVENTIONS:
Procedure: hemodiafiltration with endogenous re infusion (HFR) — hemodiafiltration with endogenous re infusion (HFR) for cases 2
  Other Names: medical treatment; Measurement of C1q levels

SUMMARY:
Background: lupus is a heterogeneous autoimmune disease with autoantibodies formation. Lupus nephritis carries the worst prognosis. C1q deficiency correlates with activity and renal involvement and may help in its evaluation. Therapies include plasma exchange, immune adsorption and recently under evaluation, hemodiafiltration with on-line endogenous re infusion (HFR), in addition to traditional immunosuppressive therapies. Aim: is to evaluate the role of HFR in improving signs and symptoms of SLE activity and laboratory parameters not responding to traditional immune suppressive therapy

DETAILED DESCRIPTION:
Settings and design: A controlled clinical study was conducted on group A, sixty patients with lupus in activity subdivided into cases 1, 47 patients, who received traditional medical treatment and cases 2 group, 13 patients, who underwent HFR in addition to medical treatment. And group B that consisted of two subgroups, control 1, 20 healthy age and sex matched volunteers and control 2, 10 cases with different glomerular diseases other than lupus.

Methods and materials: Serum c1q was done before and after the HFR as well as induction by medical treatment. Disease activity assessed using SLEDAI-2K with responder index - 50, quality of life assessed using SLEQOL v2, and HFR was performed for the non-responder group.

The study will be conducted in Alexandria University Hospitals in compliance with the Declaration of Helsinki; the ethical committee of the investigator's faculty will be requested to approve the protocol and the patients will be requested to give informed consent.

ELIGIBILITY:
Inclusion Criteria:

* systemic lupus erythematosus in activity

Exclusion Criteria:

* End stage renal disease, other renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Improvement In signs and symptoms of lupus activity assessed by Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) | 12 months
  For cases group

CONTACTS AND LOCATIONS:
Overall Officials: Naga S Salah, Professor, Principal Investigator — University of Alexandria
Locations (1):
- Faculty of Medicine Alexandria University, Alexandria, Sidi Beshr, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data will be available and can be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 2 days, forever available
Access Criteria: no specific criteria